CLINICAL TRIAL: NCT05129839
Title: The Effect of Lightened and Musical Baby Mobile on Sleep Quality in Hospitalized Children in A Pediatric Emergency Clinic: A Prospective Randomized Controlled Study
Brief Title: Use of Lightened and Musical Baby Mobile in a Pediatric Emergency Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/05-15
Record Dates: First submitted 2021-10-24; First posted 2021-11-22 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Sleep; Nursing Caries
Keywords: Pediatric emergency clinic; Sleep; Sleep quality; Lightened and musical baby mobile
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lightened and Musical Baby Mobile Group (Experimental): The children in the study group were applied a lightened and musical baby mobile before sleeping at night.
  Interventions: Device: lightened and musical baby mobile
- Control Group (No Intervention): The children in the control group were not given lightened and musical baby mobile, and their routine sleep patterns were continued.

INTERVENTIONS:
Device: lightened and musical baby mobile — Before going to sleep in the infant's room in the intervention group, a lightened and musical baby mobile was used.
  Arms: Lightened and Musical Baby Mobile Group

SUMMARY:
The aim of this study is to present results on the effect of lightened and musical baby mobile on sleep quality in children hospitalized in the pediatric emergency clinic. In the randomized controlled study, 124 children hospitalized in the pediatric emergency clinic of a public hospital and appropriate the inclusion criteria were equally divided into 2 groups. The lightened and musical baby mobile was used during the night's sleep in the patient's room of the children in the first group (intervention group). The children in the second group (control group) did not use a lightened and musical baby mobile. The sleep quality of the children in the 2 groups was evaluated with the Child's Sleep Quality Evaluation Form (CSQEF).

DETAILED DESCRIPTION:
Illness, hospital environment, hospitalization and routines; are common sources of stress experienced by children. This experience; delays the child's recovery process and growth-development, impairs play activity and sleep quality. The aim of this randomized controlled study is to present results on the effect of lightened and musical baby mobile on sleep quality in children hospitalized in the pediatric emergency clinic.

METHODS This study was conducted in a single-center, prospective randomized controlled design. The sample size of the study was calculated in the program of G* Power 3.1.9.2 (Heinrich Heine University Düsseldorf, Germany). The sample size was found to be 60 children for each group. The study authors considered possible sample losses during the study process. It was decided to conduct the study with a total of 124 children. There were 62 children in each group (intervention and control group). This study included 150 children hospitalized in a 6-bed pediatric emergency clinic of a public hospital in Istanbul between October and December 2019. Of these children, 124 children who met the inclusion criteria were included in the study. Children who were transferred to other inpatient units after hospitalization in the emergency department (n=18) and whose parents refused to participate in the study (n=8) were excluded from the study.

Procedures:

Assigning the participants to the groups, positioning and operating the lightened and musical baby mobile in the child's room, taking vital signs, collecting the data in the CSQEF and all recordings were made by the first researcher. The first researcher has 5 years of experience as a pediatric emergency nurse. In the pediatric emergency clinic, nurses work in 2 shifts (08:00-17:00 and 16:00-08:00). The first investigator works in the pediatric emergency clinic. In this study, the following procedure was applied, respectively. Each child admitted to the pediatric emergency clinic was taken to the patient's room with his mother, his clinical status was evaluated, and the children to be included in the intervention and control groups were determined. Parents of the children included in the intervention group were informed about all stages of the research process, and their verbal and written consents were obtained. Assignment of children to groups was done by simple randomization method (according to their hospitalization on odd and even number days of the calendar). Children who were hospitalized on odd-numbered days of the calendar were included in the intervention group, and children hospitalized on even-numbered days were included in the control group. For example; The child admitted to the pediatric emergency clinic on October 11 was included in the intervention group, and the child hospitalized on October 12 was included in the control group. This sequence was repeated until the number of samples was completed. In this study, all assessments were made in the same way for the children in the intervention and control groups. In this study, data on children's sleep quality and vitals signs were re-evaluated in different time periods. These time periods are: pre-intervention and intervention day. Intervention day; in the morning (at 08:00), before going to sleep (at 20:00), during sleep (at 02:00), and the next morning (at 08:00). Before the intervention; It covers between at 08:00 in the morning the day before the child is admitted to the emergency clinic and at 08:00 in the morning on the day the child is admitted to the emergency clinic. Intervention day; It covers the first day of the child's admission to the emergency clinic between at 08:00 in the morning and at 08:00 in the next day. Factors defining the sleep quality of children; It was evaluated twice, before the intervention and on the day of the intervention. Children's vital signs, intervention day; It was measured 4 times ( in the morning, before going to sleep, during sleep and the next morning), using a pulse oximetry device and an infrared thermometer. All data, except the vital signs of the children, were asked to the mothers face-to-face and their answers were recorded in the CSQEF.

Instruments:

Data were collected with the Child's Sleep Quality Evaluation Form (CSQEF). CSQEF was developed by the authors based on the literature. The questions in the form; The child's age, gender, vital signs (blood pressure, radial pulse, respiratory rate and body temperature) and factors indicating sleep quality ( night sleep duration/hour and night awakenings/number). In the study, a lightened and musical baby mobile, which facilitates the falling asleep of children and allows them to continue their sleep, was used in the rooms of the children in the hospital. In the study, In the study, a lightened and musical baby that can be hung on the wall and fixed on a flat surface was used. An illuminated musical mobile with light emitting diode (LED) lights and a reflective interior surface, providing night sky projection on the ceiling and walls, with 5 different color options, 4 function keys and soft music, was used.

Intervention:

Children in the intervention and control groups, who were admitted to the pediatric emergency clinic, were monitored by being connected to the pulse oximeter device located at the bedside. Vital signs were measured and recorded first thing in the morning (at 08:00) on the intervention day. The child's age, gender, and factors defining sleep quality before the intervention (1st evaluation) were asked face-to-face to the mothers and their answers were recorded in the CSQEF. At 19:00, a mobile with light and music was placed in the middle of the bedside table in the room of the children in the intervention group. Checked the volume, lighting color, pattern and rotation function. Sound; set to medium level, which facilitates the transition to sleep. lighting color; set to a yellow color that provides dim light and is not distracting. As a pattern; Reminiscent of the night, the moon-star projection and rotation function were used.The patient room of the children in the intervention and control groups was illuminated and the window blinds were closed to provide a dark environment. Vital signs of the children in the intervention and control groups were measured and recorded at 20:00. The mobile with light and music placed in the room of the children in the intervention group was started at 20:00. The children in the control group did not use lightened and musical baby mobile, and the routine sleep pattern was maintained. Children in the intervention and control groups at 02:00 (during sleep) and 08:00; Vital signs were measured and recorded. The next morning on the intervention day (at 08:00); The mothers in the intervention and control groups were asked face-to-face about the factors that define the sleep quality of the children in the intervention and control groups between at 20:00 and 08:00 (2nd evaluation) and that their impair (1st evaluation) and their answers were recorded in the CSQEF.

ELIGIBILITY:
Inclusion Criteria:

* Be between 1-3 years old
* Being on the 2nd day of hospitalization
* Staying with his mother in the emergency clinic for 24 hours
* Parent's consent to participate in the study
* Hospitalized due to an acute illness
* Stable clinical condition
* No painful intervention on the day of application
* No isolation
* Absence of neurological disease, mental and sensory disability

Exclusion Criteria:

* A painful procedure on the day of application
* Applying insulation
* Neurological disease
* Have a mental and sensory disability

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Identifying children's sleep quality | Change in the night sleep duration and night awakenings of children in two days.
  The child's night sleep duration (hour and minute) and night awakenings (number) were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Topsakal, Principal Investigator — Marmara Unıvesıty Educatıon And Research Hospital Pediatric Emergency Clinic Istanbul, Turkey.
Locations (1):
- Marmara Unıvesıty Educatıon And Research Hospıtal, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No